CLINICAL TRIAL: NCT03241394
Title: The Investigation of the Role of Inflammation in the Insulin Resistance Syndrome: The Monocyte Subsets in Obese Patients With and Without Metabolic Syndrome
Brief Title: The Monocyte Subsets in Obese Patients With and Without Metabolic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Ioannina (Other)
Responsible Party: Principal Investigator, Georgios A. Christou, Cardiologist, Postdoctoral researcher, University Hospital, Ioannina
Other Study IDs: 802
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: Monocyte subsets; Obesity; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lean: Individuals with Body Mass Index (BMI) = 18.5 - 25.0 Kg/m2
- Obese with MS: Individuals with BMI ≥ 30.0 Kg/m2 and metabolic syndrome (MS) MS was defined as the presence of three or more of the following criteria: 1) waist circumference ≥ 102 cm in men and ≥ 88 cm in women, 2) serum triglycerides ≥ 150 mg/dL, 3) high density lipoprotein-cholesterol (HDL-C) < 40 mg/dl in men and < 50 mg/dl in women, 4) systolic blood pressure (SBP) ≥ 130 mmHg or diastolic blood pressure (DBP) ≥ 85 mmHg or antihypertensive drug treatment, 5) fasting glucose ≥ 100 mg/dL
- Obese without MS: Individuals with BMI ≥ 30.0 Kg/m2 but not MS

SUMMARY:
Obesity is associated with a chronic low-grade inflammation characterized by macrophage infiltration in adipose tissue that induces insulin resistance and the appearance of metabolic syndrome (MS). The aim of the study was the investigation of whether circulating monocyte subsets are differentially regulated in MS.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

Age less than 18 years old, pregnancy, breast feeding, kidney disease, liver disease, gastrointestinal disease, malignancy, any endocrine disorder or metabolic disease, other than obesity or type 2 diabetes mellitus (T2DM), alteration of body weight (BW) by up of 5% of the initial BW during the last 3 months, any state of stress or systemic inflammation and taking any of the following drugs, within 3 weeks prior to the start of the study: hypolipidemic agents, antidiabetics, drugs for weight loss, nonsteroidal antiinflammatory drugs, glucocorticoids.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the present study healthy lean volunteers and obese subjects were recruited. The obese patients attended the Endocrinology outpatient clinic of the University Hospital of Ioannina in Greece. The obese patients were either with metabolic syndrome (MS) or without MS.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-07-25 (Actual); Primary Completion 2017-09-15 (Estimated); Study Completion 2017-09-15 (Estimated)

PRIMARY OUTCOMES:
Monocyte subsets | Baseline measurement
  Absolute blood count of classical (Mon1A), intermediate (Mon2A) and nonclassical (Mon3A) monocyte subsets wil be measured by flow cytometry.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Ioannina, Ioannina, Greece

REFERENCES:
- [Derived] Christou KA, Christou GA, Karamoutsios A, Vartholomatos G, Gartzonika K, Tsatsoulis A, Tigas S. Metabolically Healthy Obesity Is Characterized by a Proinflammatory Phenotype of Circulating Monocyte Subsets. Metab Syndr Relat Disord. 2019 Jun;17(5):259-265. doi: 10.1089/met.2018.0132. Epub 2019 Mar 13. PMID 30864887